CLINICAL TRIAL: NCT01961180
Title: The Effect of Cipralex in Polycystic Ovary Syndrome
Brief Title: The Effect of Cipralex on Quality of Life, Adrenal Activity Glucose Metabolism, Physical and Mental Health in PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Andersen, Professor, chief physisian, Odense University Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 24638418
Record Dates: First submitted 2013-07-03; First posted 2013-10-11 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Quality of Life; Adrenal hyper activity; Glucose metabolism
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Dexetimide; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active comparator (Active Comparator): Drug: Cipralex
  Interventions: Drug: Cipralex
- placebo comparator (Placebo Comparator): Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cipralex — the dosage is crescendo for one week and descending for two weeks with half dosage, to avoid side effects.
  Other Names: Escitalopram
  Arms: active comparator
Drug: Placebo — Placebo
  Arms: placebo comparator

SUMMARY:
Objectives: To investigate the effect of Cipralex versus placebo on stress hormones, glucose metabolism, physical and mental health and quality of life in polycystic ovary syndrome(PCOS).

Treatment: 2x20 women for 12 weeks. Design: Double blinded, randomized, placebo controlled.

DETAILED DESCRIPTION:
We want to investigate the effect of Cipralex versus placebo on stress hormones, glucose metabolism, physical and mental health and quality of life in polycystic ovary syndrome(PCOS).

PCOS is characterized by menstrual deregulation, high testosterone, mail hair growth and increased stress hormones from the adrenals. Furthermore there are changes similar to those seen in diabetes.

Cipralex is known to decrease stress hormones. But no investigations are on the effect of cipralex on PCOS, or how the increased stress hormones affect the PCOS condition.

We will examine 2x20 women with PCOS. They will be randomized to Cipralex or placebo. Treatment duration is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI >25 and <50
* Age < 50
* PCOS

Exclusion Criteria:

* Epilepsia
* use of metformin or oral anticonceptives
* pregnancy/breastfeeding

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-06; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 14 weeks
  Measured by questionaires

SECONDARY OUTCOMES:
Level of cortisone in 24 hour urine sample | June 2013 to October 2015
  Cortisone and cortisone metabolites, measured by 24 hour urine sample.

OTHER OUTCOMES:
Glucose metabolism | June 2013 to October 2015
  measures bu 3 hour Glucose Tolerance Test, and homeostasis model assessment-insulin resistance(HOMA-IR)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne MD Andersen, sponsor, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Endocrinology, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes